CLINICAL TRIAL: NCT00214565
Title: A 24-Wk Randomised, Double-Blind, Multi-Centre, Active-Controlled (Pioglitazone) Study to Evaluate the Efficacy, Safety & Tolerability of Tesaglitazar Therapy When Administered to Patients With Type 2 Diabetes
Brief Title: GALLANT 6 Tesaglitazar vs. Pioglitazone
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The development program has been terminated
Sponsor: AstraZeneca (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D6160C00030
Record Dates: First submitted 2005-09-20; First posted 2005-09-22 (Estimated); Last update posted 2010-11-19 (Estimated); Status verified 2010-11

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Type 2 diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — tesaglitazar

INTERVENTIONS:
Drug: Galida

SUMMARY:
This is a 24-week randomized, double-blind, multi-center, active-controlled (pioglitazone) study of tesaglitazar (0.5 mg and 1 mg) in patients with type 2 diabetes, not adequately controlled on diet and lifestyle advice alone during the run-in period. The study comprises a 3-week enrollment period, 6 week placebo single blind run in period followed by a 24-week double blind treatment period and a 3-week follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Provision of a written informed consent
* Men or women who are ³18 years of age
* Female patients: postmenopausal, hysterectomized, or if of childbearing potential, using a reliable method of birth control
* Diagnosed with type 2 diabetes
* Treated with diet alone or treatment with a single oral antidiabetic agent or low doses of two oral antidiabetic agents

Exclusion Criteria:

* Type 1 diabetes
* New York Heart Association heart failure Class III or IV
* Treatment with chronic insulin
* History of hypersensitivity or intolerance to any peroxisome proliferator-activated receptor agonist (like Actos or Avandia), fenofibrate, metformin or 3-hydroxy-3-methylglutaryl coenzyme A reductase inhibitor (statin)
* History of drug-induced myopathy or drug-induced creatine kinase elevation, liver enzyme elevations, neutropenia (low white blood cells)
* Creatinine levels above twice the normal range
* Creatine kinase above 3 times the upper limit of normal
* Received any investigational product in other clinical studies within 12 weeks
* Any clinically significant abnormality identified on physical examination, laboratory tests or electrocardiogram, which in the judgment of the investigator would compromise the patient's safety or successful participation in the clinical study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1450
Dates: Start 2004-08; Primary Completion 2006-10 (Actual); Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
Absolute change from baseline to end of randomized treatment period in glycosylated hemoglobin A1c (HbA1c)

SECONDARY OUTCOMES:
The change in fasting plasma glucose (FPG), insulin, proinsulin and C-peptide
Insulin sensitivity by assessment of change in the calculated variable homeostasis assessment model
Lipid parameters
FPG, homeostasis assessment model, insulin, proinsulin, C-peptide
Responder analyses for HbA1c, FPG, TG, HDL C, total cholesterol, non HDL C and LDL C according to pre-specified values
Pharmacokinetics of tesaglitazar
Safety and tolerability of tesaglitazar by assessment of adverse events, laboratory values, electrocardiogram, pulse, blood pressure, hypoglycemic events, body weight, cardiac evaluation, and physical examination
Assess the effects on patient-reported outcomes using the Medical Outcomes Study Short Form-36 (SF-36)
Validate the Work Productivity and Activity Impairment-Diabetes Questionnaire (WPAI Diabetes) and the Diabetes Productivity Impairment Questionnaire (DPIQ) (US only).

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca Galida Medical Science Director, MD, Study Director — AstraZeneca
Locations (74):
- Research Site, Altoona, Pennsylvania, United States
- Argentina (6):
  - Research Site, Ciudad de Buenos Aires
  - Research Site, Córdoba
  - Research Site, Moron- Buenos Aires
  - Research Sites, Quilmes - Buenos Aires
  - Research Site, Rosario
  - Research Site, Salta
- Research Site, Curitiba, Brazil
- Canada (23):
  - Research Site, Edmonton, Alberta
  - Research Site, Abbotsford, British Columbia
  - Research Site, Chilliwack, British Columbia
  - Research Site, Vancouver, British Columbia
  - Research Site, Victoria, British Columbia
  - Research Site, Dartmouth, Nova Scotia
  - Research Site, Halifax, Nova Scotia
  - Research Site, Truro, Nova Scotia
  - Research Site, Windsor, Nova Scotia
  - Research Site, Brampton, Ontario
  - Research Site, Etobicoke, Ontario
  - Research Site, Kingston, Ontario
  - Research Site, Niagara Falls, Ontario
  - Research Site, Oshawa, Ontario
  - Research Site, Scarborough Village, Ontario
  - Research Site, St. Catharines, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Windsor, Ontario
  - Research Site, Trois-Rivières, Quebec
  - Research Site, Chicoutimi
  - Research Site, Longueuil
  - Research Site, Montreal
  - Research Site, St. John's
- Finland (6):
  - Research Site, Espoo
  - Research Site, Helsinki
  - Research Site, Kuopio
  - Research Site, Pietarsaar
  - Research Site, Pori
  - Research Site, Tampere
- Mexico (7):
  - Research Site, Guadalajara Jalisco
  - Research Site, Mexico City
  - Research Site, México
  - Research Site, Nuevo León
  - Research Site, Puebla City
  - Research Site, Torreón
  - Research Site, Zapopan
- Norway (15):
  - Research Site, Ås
  - Research Site, Bergen
  - Research Site, Elvernum
  - Research Site, Hamar
  - Research Site, Horten
  - Research Site, Kongsberg
  - Research Site, Lena
  - Research Site, Loeten
  - Research Site, Lysaker
  - Research Site, Oslo
  - Research Site, Osteraas
  - Research Site, Skedsmokorset
  - Research Site, Straume
  - Research Site, Tronheim
  - Research Site, Tønsberg
- United Kingdom (15):
  - Research Site, Dublin, Ireland
  - Research Site, Wexford, Ireland
  - Research Site, Antrim, NI
  - Research Site, Belfast
  - Research Site, Cardiff
  - Research Site, Edinburgh
  - Research Site, Glasgow
  - Research Site, Kent
  - Research Site, Leeds
  - Research Site, Mid Glamorgan
  - Research Site, Pembrokeshire
  - Research Site, Plymouth
  - Research SIte, Reading
  - Research Site, Surrey
  - Research Site, Wiltshire